CLINICAL TRIAL: NCT01181388
Title: Impacts of Superselective Infarct-related Artery Infusion of Tirofiban on Myocardial Reperfusion and Bleeding Complications in ST Segment Elevation Myocardial Infarction (STEMI) Patients
Brief Title: Impacts of Superselective Infarct-related Artery (IRA) Infusion of Tirofiban on Myocardial Reperfusion and Bleeding Complications in Acute Myocardial Infarction (AMI) Patients
Acronym: SUIT-AMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Hongbing Yan, the 28th Division, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 64456541
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2010-06

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

ARMS (2):
- intra-guide-catheter infusion of tirofiban (Active Comparator)
  Interventions: Procedure: administration of tirofiban by guide catheter
- intra-thrombus-aspiration-catheter infusion of tirofiban (Experimental)
  Interventions: Procedure: administration of tirofiban by thrombus aspiration catheter in infarct-related artery

INTERVENTIONS:
Procedure: administration of tirofiban by thrombus aspiration catheter in infarct-related artery — a bolus of 10ug/kg tirofiban administration via thrombus aspiration catheter followed by 0.1ug/kg/min for 12 hours after PCI
  Arms: intra-thrombus-aspiration-catheter infusion of tirofiban
Procedure: administration of tirofiban by guide catheter — a bolus of 10ug/kg tirofiban administration via guide catheter followed by 0.1ug/kg/min for 12 hours after PCI
  Arms: intra-guide-catheter infusion of tirofiban

SUMMARY:
Superselective IRA infusion of tirofiban may improve myocardial reperfusion and reduce bleeding complications in AMI patients.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients
* chest pain for less than 12hr
* plan to PCI

Exclusion Criteria:

* LM lesion
* stent thrombosis
* cardiac shock
* thrombocytopenia
* allergy to asprin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 1 month after PCI
  Infarct size, reinfarction, motality, et.al.
Major adverse cardiovascular events | 3 months after PCI
  Infarct size, reinfarction, motality, et.al.
Major Adverse Cardiovascular Events | 6 months after PCI
  Infarct size, reinfarction, motality, et.al.

SECONDARY OUTCOMES:
number of participants with bleeding events | 1 month
  bleeding events are assessed by Thrombolysis In Myocardial Infarction(TIMI) criteria

CONTACTS AND LOCATIONS:
Locations (1):
- the 28th division, Beijing Anzhen Hospital, Beijing, Beijing Municipality, China